CLINICAL TRIAL: NCT04164173
Title: Hyperinflation Respiratory Therapies in Cardiac Surgery Patients: A Randomized, Observer-Blinded, Prospective Clinical Trial
Brief Title: Hyperinflation Respiratory Therapies in Cardiac Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jaffer Odeh, Assistant Profesor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU-2019-1242
Record Dates: First submitted 2019-11-08; First posted 2019-11-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease; Postoperative Complications
MeSH Terms: conditions — Lung Diseases; Postoperative Complications | interventions — Intermittent Positive-Pressure Breathing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment respiratory therapist will be blinded to respiratory therapy modalities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- EzPAP (Experimental): The patient will have EzPAP postoperative respiratory therapy as 3 x 10 breaths at a 1:4 ratio four times daily
  Interventions: Device: EzPAP
- Metaneb (Experimental): The patient will have Metaneb postoperative respiratory therapy as 10 minutes Continuous Positive End Expiratory Pressure (CPEP) four times daily
  Interventions: Device: Metaneb
- Intermittent Positive Pressure Breathing (IPPB) (Experimental): The patient will have Intermittent positive pressure breathing (IPPB) postoperatively for 10 minutes four times daily
  Interventions: Device: Intermittent Positive Pressure Breathing (IPPB)

INTERVENTIONS:
Device: EzPAP — Patient will receive 10 min EzPAP 4 times daily
  Other Names: Postoperative hyperinflation therapy-EzPAP
  Arms: EzPAP
Device: Metaneb — Patient will receive 10 min Metaneb 4 times daily
  Other Names: Postoperative hyperinflation therapy-Metaneb
  Arms: Metaneb
Device: Intermittent Positive Pressure Breathing (IPPB) — Patient will receive 10 min IPPB 4 times daily
  Other Names: Postoperative hyperinflation therapy-IPPB
  Arms: Intermittent Positive Pressure Breathing (IPPB)

SUMMARY:
The purpose of this prospective randomized clinical trial is to evaluate three different types of hyperinflation respiratory therapies, Intermittent Positive Pressure Breathing (IPPB), Intermittent positive end expiratory pressure (EzPAP), Metaneb. Investigators will examine which hyperinflation therapy provides better lung expansion and may improve lung recovery after surgery.

DETAILED DESCRIPTION:
Postoperative pain due to surgical incision may limit lung expansion. After cardiac surgery, all patients receive respiratory therapies, because it is critical to expand lung after surgery to prevent respiratory complications such as lung collapse (atelectasis) due to shallow breathing or accumulation of airway secretions.

Although incentive spirometer is the most common method used for lung recovery after cardiac surgery, some studies were not able to find any benefits from the use of incentive spirometer. Inspiratory positive-pressure breathing (IPPB), Intermittent positive end expiratory pressure (EzPAP), and chest airway clearance (Metaneb) are hyperinflation therapies used after surgery. The purpose of this research study is to determine which hyperinflation respiratory therapy provide better lung recovery after cardiac surgery.

Hyperinflation Respiratory Therapies:Participants will be randomly assigned one of the hyperinflation respiratory therapy, intermittent positive pressure breathing (IPPB) and the EzPAP or the Metaneb.

1. Intermittent positive pressure breathing (IPPB) is a respiratory therapy technique which will support your breathing by providing pressure support. This respiratory method will increase air volume breathing in.
2. The EzPAP is another respiratory treatment and participants will breath against to resistance in order to prolong the time the lung remain open.
3. The Metaneb will provide resistance when patients breathing in order to prolong the lung opening.

Hyperinflation therapy will be performed every 4 hours in the intensive care unit (ICU). Each respiratory therapy session will take about 15 minutes. Participants' pulmonary function will be evaluated daily to monitor the lung recovery with microspirometer which will take place approximately 5 minutes. Total study duration is about 96 hours after surgery or until discharge from the Intensive Care Unit.

Risk for Lung over expansion (hyperinflation) therapy:

Hyperinflation respiratory treatments target to expand your lung to prevent complication such as collapse of small airway after surgery. This over expansion of your lung may increase work of breathing. All expected complications are typical in the post-operative cardiac patients and not unique to hyperinflation therapy.

The possible complications listed below:

1. Over distention of air sucks (alveoli). Sometimes pressure trauma in your lung may cause pneumothorax.
2. Infection
3. Bloody sputum (hemoptysis)
4. Blood gas changes such as decrease carbon dioxide or increase oxygen in your blood.
5. Sometimes stomach may distend
6. Impaction of airway secretions if gas mixture not humidified enough.
7. Your blood return to the heart maybe decreased which may affect your blood pressure.
8. Exacerbation of low blood oxygen level (hypoxemia),
9. Decreased or increased respiration
10. Air trapping in your airway
11. You may psychologically dependence to device

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Admitted to Cardiovascular ICU (CVICU) after coronary artery bypass grafting (CABG), isolated valve repair/replacement, or CABG + valve repair/replacement
3. Cardiac surgery performed via median sternotomy

Exclusion Criteria:

1. BMI>40
2. Refusal to be consented
3. Prior or current lung transplant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative lung function as assessed by the changes in FEV1/FVC | Up to 96 hours postoperatively or until discharge from the intensive care unit (ICU), whichever came first.
  The postoperative changes in the Forced Expiratory Volume in one second (FEV1)/the Forced Vital Capacity (FVC) in microspirometry

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Odeh, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Clements University Hospital, Dallas, Texas, United States